CLINICAL TRIAL: NCT02748707
Title: Effect of COX-2 (Cyclooxygenase-2) and EGFR (Epidermal Growth Factor Receptor) Suppression on Molecular Markers of Angiogenesis and Proliferation in Squamous Cell Carcinoma of Oral Cavity - Prospective Randomized Study.
Brief Title: Effect of COX-2 and EGFR Suppression on Molecular Markers of Angiogenesis and Proliferation in Squamous Cell Carcinoma of Oral Cavity - Prospective Randomized Study
Acronym: ERLO-XIB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Sudhir Nair, Associate Professor, Tata Memorial Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 830
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Oral Squamous Cell Carcinoma; Carcinoma of Buccal Mucosa; Tongue Cancers; Head and Neck Cancers
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms; Head and Neck Neoplasms | interventions — 26S proteasome non-ATPase regulatory subunit 13; Celecoxib; DMAC2L protein, human; Erlotinib Hydrochloride; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental): Celecoxib 200mg twice daily for 21 days
  Interventions: Drug: Arm1
- Arm 2 (Experimental): Erlotinib 150 mg once daily for 21 days
  Interventions: Drug: Arm 2
- Arm 3 (Experimental): Celecoxib 200 mg twice daily for 21 days and Erlotinib 150 mg once daily for 21 days
  Interventions: Drug: Arm 3
- Arm 4 (Sham Comparator): Control group with no drug
  Interventions: Other: Arm 4

INTERVENTIONS:
Drug: Arm1 — Drug (Celecoxib as 200mg twice daily) given orally for 21 days after confirmation by biopsy and before definitive treatment by surgery
  Other Names: Celecoxib
  Arms: Arm 1
Drug: Arm 2 — Drug (ERLOTINIB 150 mg daily) given orally for 21 days after confirmation by biopsy and before definitive treatment by surgery
  Other Names: Erlotinib
  Arms: Arm 2
Drug: Arm 3 — Drugs (Celecoxib 200mg twice daily and Erlotinib 150mg once daily) given orally for 21 days after confirmation by biopsy and before definitive treatment by surgery
  Other Names: Celecoxib + Erlotinib
  Arms: Arm 3
Other: Arm 4 — Patients randomized to this arm will be observed for 21 days before definitive treatment by surgery.Having a control group is ethically justifiable because the average waiting time in our hospital prior to definitive treatment is 30 days after diagnosis.
  Other Names: Observation
  Arms: Arm 4

SUMMARY:
This is a phase II randomized clinical trial to study the effect of COX-2 inhibitor Celecoxib and EGFR tyrosine kinase inhibitor Erlotinib alone or in combination on molecular markers of apoptosis and angiogenesis.

DETAILED DESCRIPTION:
Activation of EGFR signalling can lead to increased transcription of COX-2. Increased COX-2 transcription results in enhanced production of PGs, including PGE2, which in turn can activate EGFR initiating a positive feedback loop. Although majority of HNSCC over-express EGFR, the clinical responses to EGFR targeting agents have been modest. When the mechanisms of intrinsic resistance are identified like the mutations in the EGFR receptor, alternative therapeutic approaches should be employed. In preclinical studies, combining an inhibitor of COX-2 with an inhibitor of EGFR tyrosine kinase was more effective than either agent alone in suppressing tumor formation. Acquired resistances that may be amenable to pharmacological intervention include deregulation of EGFR degradation, constitutive activation of overlapping signal transduction pathways, especially cMET/HER3, the PI3K/Akt resistance pathway, angiogenesis and epithelial to mesenchymal transition. Preclinical data suggest that COX-2 inhibitors can affect most of the described acquired EGFR resistance pathways.

We propose a prospective phase II randomized trial based on a 2 X 2 factorial design in which patients are randomized to COX-2 inhibition vs. no COX-2 inhibition. Each arm will be further randomized to erlotinib vs. no erlotinib. This results in the following treatment combinations.

Arm 1: Celecoxib 200mg twice daily Arm 2: Celecoxib 200mg twice daily + Erlotinib 150mg daily Arm 3: Erlotinib 150mg alone Arm 4: Control group with no drug Patients in the drug treatment arm will receive the prescribed drug for 21 days before the tumor being surgically resected. Having a control group is ethically justifiable because the average waiting time in our hospital prior to definitive treatment is 30 days after diagnosis.

The study population consists of any patients with resectable oral cavity squamous cell carcinoma seen at Tata memorial hospital. Tumor size will be estimated by MRI Scans as well as by clinical examination before and after completion of the study drugs.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with squamous cell carcinoma of oral cavity (T2-T4, N1-2, M0) and are candidates for first line curative surgical treatment and are able to swallow orally, preoperatively.
2. Patients must be at least 18 years of age.
3. All patients must sign an informed consent before enrolling in study.
4. Patients must be able and willing to return to the clinic at appropriately scheduled intervals.
5. No use of systemic steroids or topical oral steroid preparations within three months. (Topical nasal steroid sprays or cutaneous preparations with minimal systemic absorption for nasal or dermatologic disorders are allowed).
6. Premenopausal women must be using adequate birth control methods and have a negative pregnancy test prior to entry.
7. Karnofsky Performance Score above 80.
8. The subject is willing and able to fully participate for the duration of the study.
9. If applicable, the subject has been counseled on smoking cessation.
10. The subject meets the following laboratory eligibility criteria during a time not to exceed 4 weeks prior to randomization.
11. Hemoglobin level above 10gm/dl, the lower limit of normal.
12. WBC count > 3,000 mm3.
13. Platelets count > 100,000 m3.
14. Total bilirubin, AST (Aspartate Aminotransferase) and ALT (Alanine transaminase) ≤ 2 x ULN.
15. Serum creatinine ≤ 2 x Upper limit of Normal (ULN)

Exclusion Criteria:

1. History of cardiovascular co morbidities 2. Patients with previous history of head and neck cancers 3. Recent massive gastrointestinal hemorrhage 4. An on-going unmanaged serious infectious disease or major metabolic disorder 5. Neutrophil count of <1 x 109 per liter or platelet count of < 75 x 109 per liter at study entry, 6. Bilirubin at >1.5-fold above the upper limit of normal, and 7. Kidney failure (Glomerular filtration rate of <40 mL/min). 8. Pregnant women 9. Use other nonsteroidal anti-inflammatory drugs (NSAIDs) or corticosteroids within 2 weeks prior to initial clinical evaluation 10. The subject is, in the opinion of the Institutional Principal Investigator, not an appropriate candidate for study participation.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in expression of selected biomarkers in tissue samples, assessed by immunohistochemistry (IHC) and PCR | baseline and 21 days
  Tumor tissues will be collected and stored before and after treatment. The pre and post treatment tumor tissue will be analyzed semiquantitatively by immunohistochemistry for the levels of COX-2 (Cyclooxygenase-2), EGFR (epidermal growth factor receptor), TP53 (Tumor protein 53) and VEGF (Vascular endothelial growth factor) expression. Their baseline gene expression and fold change after treatment will be assessed by quantitative real time polymerase chain reaction (qPCR) using facility at TMC.

SECONDARY OUTCOMES:
Clinical and radiological Change in tumor size and appearance | baseline and 21 days

OTHER OUTCOMES:
Disease free survival | Date of randomization to date of disease recurrence, or appearance of a new primary or death.

CONTACTS AND LOCATIONS:
Overall Officials: Sudhir V Nair, MBBS, MS,MCh, Principal Investigator — Tata Memorial Center
Locations (1):
- Tata Memorial Center (TMC), Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No